CLINICAL TRIAL: NCT01794832
Title: A Prospective Longitudinal Study of Severe Aortic Stenosis in Elderly and Outcome of Aortic Surgery.
Brief Title: Severe Aortic Stenosis in Patients Referred for Valve Surgery
Acronym: SAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Amjad Iqbal Hussain, Md, Oslo University Hospital
Other Study IDs: SAS
Record Dates: First submitted 2013-02-16; First posted 2013-02-20 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Aortic Stenosis; Valvular Heart Disease; Symptomatic Aortic Stenosis
Keywords: HRQoL; Aortic stenosis; Aortic valve surgery
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Serum, myocardial biopsi
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly with severe aortic stenosis: Patients with severe symptomatic aortic stenosis referred for consideration of surgical aortic valve replacement

SUMMARY:
Our main hypothesis on the present study is that new parameters such as risk-taking behavior, patients motivation, health related quality of life, new biomarkers and more precise echocardiography measures in addition to traditional parameters will improve pre-operative risk assessment in patients with AS and better guide patients and doctors in decision whether to operate or not.

DETAILED DESCRIPTION:
Patients referred for surgery are included thorough reading referral letter. Data collected in the study wil be compared with data from Medical records and clinical examination.

Data entered will be controlled by two investigators.

Data wil be compared to national norms and from result of other studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years with symptomatic AS referred to preoperative examination.

Exclusion Criteria:

* Exclusion: Patients who do not want to participate. Patients not able to speak and read Norwegian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion: Patients above 18 years with symptomatic AS referred to preoperative examination will be included. Patients will undergo standard investigations with regard to assessment of the clinical indication for operation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-02; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Death due cardiovascular events | one year

SECONDARY OUTCOMES:
MACE ( Major cardiovascular events ) | 30 days
  Cerebral complications (stroke/bleeding), bleeding, renal failure, arrythmias, needs for pacemaker, prolong ICU stay, wound infections

OTHER OUTCOMES:
Change in Health related Quality and function one year after inclusion | one year
  Patients in the study perform Short Form-36, EuroQual-5D at inclusion and one year after. We want to compare the result of their scoring to obtain the gain in HRQoL of the intervention
Hospital visit and use of Health services last years | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kjell I Pettersen, MD, Study Director — University of Oslo; Amjad I Hussain, MD, Principal Investigator — Oslo University Hosptial; Lars Gullestad, Professor, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University hospital- Rikshospitalet, Oslo, Norway

REFERENCES:
- [Derived] Arain F, Abraityte A, Bogdanova M, Solberg OG, Michelsen AE, Lekva T, Aakhus S, Holm S, Halvorsen B, Finsen AV, Vinge LE, Nymo S, Espeland T, Ranheim T, Aukrust P, Vaage IJ, Auensen A, Gullestad L, Ueland T. YKL-40 (Chitinase-3-Like Protein 1) Serum Levels in Aortic Stenosis. Circ Heart Fail. 2020 Oct;13(10):e006643. doi: 10.1161/CIRCHEARTFAILURE.119.006643. Epub 2020 Sep 23. PMID 32962417
- [Derived] Kvaslerud AB, Hussain AI, Auensen A, Ueland T, Michelsen AE, Pettersen KI, Aukrust P, Morkrid L, Gullestad L, Broch K. Prevalence and prognostic implication of iron deficiency and anaemia in patients with severe aortic stenosis. Open Heart. 2018 Dec 16;5(2):e000901. doi: 10.1136/openhrt-2018-000901. eCollection 2018. PMID 30613413
- [Derived] Hussain AI, Auensen A, Brunborg C, Beitnes JO, Gullestad L, Pettersen KI. Age-dependent morbidity and mortality outcomes after surgical aortic valve replacement. Interact Cardiovasc Thorac Surg. 2018 Nov 1;27(5):650-656. doi: 10.1093/icvts/ivy154. PMID 29746650
- [Derived] Auensen A, Hussain AI, Garratt AM, Gullestad LL, Pettersen KI. Patient-reported outcomes after referral for possible valve replacement in patients with severe aortic stenosis. Eur J Cardiothorac Surg. 2018 Jan 1;53(1):129-135. doi: 10.1093/ejcts/ezx228. PMID 28977361
- [Derived] Hussain AI, Garratt AM, Brunborg C, Aakhus S, Gullestad L, Pettersen KI. Eliciting Patient Risk Willingness in Clinical Consultations as a Means of Improving Decision-Making of Aortic Valve Replacement. J Am Heart Assoc. 2016 Mar 18;5(3):e002828. doi: 10.1161/JAHA.115.002828. PMID 26994130